CLINICAL TRIAL: NCT00650039
Title: A Multicenter, Double-Blind, Placebo-Controlled, Randomized Study Of The Analgesic Efficacy And Safety Of Valdecoxib 20 Mg QD And Valdecoxib 20 Mg BID Compared To Placebo Over Multiple Days For Management Of Acute Postsurgical Pain In Patients Undergoing Anterior Cruciate Ligament Reconstruction
Brief Title: Double-Blind, Randomized Study Of The Analgesic Efficacy And Safety Of Valdecoxib 20 Mg Daily And Valdecoxib 20 Mg Twice Daily Compared To Placebo For Management Of Acute Postsurgical Pain In Anterior Cruciate Ligament (ACL) Reconstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3471109
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-03

CONDITIONS: Pain
Keywords: Post surgical pain; Anterior Cruciate ligament reconstruction; Arthroscopy; Perioperative pain
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — valdecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 2 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — valdecoxib 40 mg (two 20-mg tablets) by mouth followed by valdecoxib 20 mg 1 to 12 hours after the first dose or 12 hours after the first dose, but no later than midnight on Day 1; then, placebo BID by mouth on Days 2 to 5.
  Arms: Arm 3
Drug: valdecoxib — valdecoxib 40 mg (two 20-mg tablets) by mouth followed by valdecoxib 20 mg 1 to 12 hours after the first dose or 12 hours after the first dose, but no later than midnight on Day 1; then, valdecoxib 20 mg once daily (QD) by mouth on Days 2 to 5.
  Arms: Arm 2
Drug: valdecoxib — valdecoxib 40 mg (two 20-mg tablets) by mouth followed by valdecoxib 20 mg 1 to 12 hours after the first dose or 12 hours after the first dose, but no later than midnight on Day 1; then, valdecoxib 20 mg twice daily (BID) by mouth on Days 2 to 5.
  Arms: Arm 1

SUMMARY:
The primary objective was to evaluate the analgesic efficacy of valdecoxib 20 mg daily and valdecoxib 20 mg twice daily compared with placebo in outpatients with moderate-severe pain after arthroscopic anterior cruciate ligament (ACL) reconstruction surgery. Secondary objectives were to compare each valdecoxib dose with placebo on additional measures of pain intensity, health outcomes, the use of rescue medication, and the occurrence of opioid-related symptoms, and to evaluate their safety.

ELIGIBILITY:
Inclusion Criteria:

* Included patients had uncomplicated arthroscopic ACL reconstruction
* Subjects were to have a Baseline pain intensity of ≥ 50 mm as measured on a 0 - 100mm visual analogue scale (VAS) and moderate to severe pain on a categorical scale by 23:00 hours on the day of surgery and prior to being discharged from the surgical facility
* Subjects could not have received any medication or additional procedures that would confound the interpretation of the study results.

Exclusion Criteria:

* the patient was admitted to or retained in the surgical center/hospital for >23 hours;
* the patient underwent any other surgical procedure, along with the orthopedic procedure, that was expected to produce a greater degree of surgical trauma than the orthopedic procedure alone;
* the patient used conventional nonsteroidal antiinflammatory drugs (NSAIDs), selective cyclooxygenase-2 (COX-2) inhibitors, or tramadol during the 6 hours preceding surgery, during surgery, or subsequent to the end of surgery;
* the patient received oxaprozin or piroxicam within 1 week prior to randomization;
* the patient had a pain pump or indwelling catheter during surgery that administered local or intraarticular anesthetics or narcotics at the index joint, or had such an intra-articular injection at the end of surgery;
* the patient had been treated with patient-controlled analgesia or NSAIDs subsequent to the end of anesthesia;
* patient had a history of clinically significant GI disease or renal disease, or history of a gastrointestinal ulcer, or cancer, or a laboratory abnormality that would suggest it was not in the subject's best interest to enroll in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2004-03; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Summed Pain Intensity (categorical) through 24 hours (SPI 24) | Day 2 and Day 3
Patient's Global Evaluation of Study Medication (PGESM) | Day 2 and Day 3

SECONDARY OUTCOMES:
Average Pain Intensity (derived from the mBPI-sf) on each study day | Days 2 to 5
Worst Pain Intensity (derived from the Modified Brief Pain Inventory Short Form [mBPI-sf]) on each study day | Days 2 to 5
Symptom Distress Scale Questionnaire | Days 2 to 5
Patient Satisfaction Questionnaire for each study day | Days 2 to 5
Time-specific pain intensity (PI) (categorical) on each study day | Days 2 to 5
SPI 24 (Visual Analog Scale [VAS]) on each study day | Days 2 to 5
Time-specific PI (VAS) on each study day | Days 2 to 5
Patient's Global Evaluation of Study Medication | Day 4 and Day 5
Time to first dose of rescue medication (supplemental analgesia) on each study day | Days 2 to 5
Percent of subjects who took rescue medication (supplemental analgesia) on each study day | Days 2 to 5
Amount of rescue medication (supplemental analgesia) taken on each study day | Days 2 to 5
Individual and Composite Pain Interference With Function score (derived from the mBPI-sf) on each day | Days 2 to 5
Time between doses of study medication on each study day | Days 2 to 5
Post-Discharge Recovery Experience for each study day | Days 2 to 5
SPI 24 (categorical) | Day 4 and Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (56):
- United States (49):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Northport, Alabama
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Pheonix, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tempe, Arizona
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, Laguna Hills, California
  - Pfizer Investigational Site, Laguna Woods, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Avon, Connecticut
  - Pfizer Investigational Site, Cromwell, Connecticut
  - Pfizer Investigational Site, Enfield, Connecticut
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, Glastonbury, Connecticut
  - Pfizer Investigational Site, Hartford, Connecticut
  - Pfizer Investigational Site, Rocky Hill, Connecticut
  - Pfizer Investigational Site, Windsor, Connecticut
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, Saint Augustine, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Weston, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Morrow, Georgia
  - Pfizer Investigational Site, Stockbridge, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Oak Park, Illinois
  - Pfizer Investigational Site, Cedar Rapids, Iowa
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Timonium, Maryland
  - Pfizer Investigational Site, Royal Oak, Michigan
  - Pfizer Investigational Site, Troy, Michigan
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Bend, Oregon
  - Pfizer Investigational Site, Anderson, South Carolina
  - Pfizer Investigational Site, Cola, South Carolina
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Orangeburg, South Carolina
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, San Marcos, Texas
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Fairfax, Virginia
- Canada (7):
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Ajax, Ontario
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, Scarborough Village, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Weston, Ontario

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3471109&StudyName=Double-Blind%2C%20Randomized%20Study%20Of%20The%20Analgesic%20Efficacy%20And%20Safety%20Of%20Valdecoxib%2020%20Mg%20Daily%20And%20Valdecoxib%2020%20Mg%20Twice%20Daily%20Compa